CLINICAL TRIAL: NCT04072965
Title: Cross Education Effect of Balance Program in Patients With Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nadia Magdy Amen Elsotohy, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cross Education of balance
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Balance; Ankle Instability

STUDY DESIGN:
Intervention Model Description: group (A) Cross Education group(B) Traditional training group (C) control
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cross eduacation of balance (Experimental): 10 females with Chronic Ankle Instability will receive balance training for the non affected side for a six weeks
  Interventions: Other: balance training
- Traditional training (Experimental): 10 females with Chronic Ankle Instability will receive balance training for the affected side for a six weeks
  Interventions: Other: balance training
- control (No Intervention): balance of 15 females with Chronic Ankle Instability will be assessed before and after six weeks of no intervention

INTERVENTIONS:
Other: balance training — Thirty five females with CAI will be recruited from the Faculty of Physical Therapy, Cairo University by announcements to participate in this study. The participants will be randomly assigned into three groups; (A) Cross Education will receive single leg balance training for the non affected side (n=10), (B) Traditional training will receive single leg balance training for the affected side (n=10), (C) control group will receive no intervention (n=15).
  Arms: Cross eduacation of balance; Traditional training

SUMMARY:
Researchers recommended that NeuroMuscularControl (NMC) training should not begin immediately after an acute Lateral Ankle Sprain(LAS) because of pain and weight-bearing restrictions. So, there is a need for an alternative way by which we can begin NMC retraining sooner. By training the non-affected ankle (Cross education), clinicians can begin NMC retraining before the individuals can bear weight on the affected ankle, in the acute stage of healing, or even if there is any other precautions or contraindications to exercise due to the injuries. Athletes with more chronic injuries may be able to perform NMC and functional retraining at higher levels than otherwise would be possible by initiating the training on the non affected ankle. Initiating these activities on the non-affected ankle will result in earlier improvements in postural control and function in the affected ankle.

By this way, the rehabilitation times will be short, athletes can return earlier to sport participation or work, health care costs will decrease. Up to the knowledge of the author, there is a gap in research investigating cross education effect of balance program in patients with ankle instability. So, the current study was conducted to reveal the role of this phenomena in such cases and add this phenomenon on the physical therapy field to manage patients with ankle instability (If Cross Education phenomena is effective, this phenomena will be used in rehabilitation).

DETAILED DESCRIPTION:
Thirty five females with Chronic Ankle Instability will be recruited from the Faculty of Physical Therapy, Cairo University by announcements to participate in this study. They will be randomly assigned into three groups; (A) Cross Education (balance training for the non affected side )(n=10), (B) Traditional training(balance training for the affected side) (n=10), (C) control group (no intervention) (n=15). stability indices measured by the Biodex Balance system , Single Leg Stance Test and scores of Star Excursion Balance Test will be assesssed before and after six weeks of Single Leg Balance training.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 ankle sprain, with the initial sprain occurring more than 1 year before the study
* A feeling of ''giving way'' (at least 2 episodes in the 6 months before the study).
* At least two ''yes'' answers on questions four to eight on the Modified Ankle Instability Instrument (MAII)

Exclusion Criteria:

1. - A history of previous surgeries or fractures in either limb of the lower extremities.
2. - Acute injury to musculoskeletal structures of other joints of the lower extremity in the previous three months, which impacted joint integrity and function (ie, sprains, fractures) resulting in at least one interrupted day of desired physical activity.
3. - Balance deficits due to vestibular disorders, such as vertebrabasilar insufficiency and/or visual disorders.
4. - Neuropathies and diabetes

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-23 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Assessing change in the Anterior reach distance of Star excursion balance test between the initial assessment and after six weeks of single leg balance training | 6 weeks
  The maximum distance the patient is able to reach in the Anterior direction during standing on one leg measured by centimeter
Assessing change in the Posteromedial reach distance of Star excursion balance test between the initial assessment and after six weeks of single leg balance training | 6 weeks
  The maximum distance the patient is able to reach in the Posteromedial direction during standing on one leg measured by centimeter
Assessing change in the Posterolateral reach distance of Star excursion balance test between the initial assessment and after six weeks of single leg balance training | 6 weeks
  The maximum distance the patient is able to reach in the Posterolateral direction during standing on one leg measured by centimeter
Assessing change in the Composite reach distance of Star excursion balance test between the initial assessment and after six weeks of single leg balance training | 6 weeks
  The mean of the anterior,Posteromedial and Posterolateral reach distances will be divided by the three times the limb lenght of the each patient
Assessing change in the Medio-lateral Stability Index (MLSI) measured by the Biodex Balance system between the initial assessment and after six weeks of single leg balance training | 6 weeks
  The Medio-lateral Stability Index (MLSI) assess the fluctuations from the horizontal along Medio-Lateral (ML) axis of the Biodex Balance System
Assessing change in the Antero-posterior Stability Index (APSI) measured by the Biodex Balance System between the initial assessment and after six weeks of single leg balance training | 6 weeks
  The Antero-posterior Stability Index (APSI) assess the fluctuations from the horizontal along the Antero-Posterior (AP) axis of the BBS
Assessing change in the Overall Stability Index (OASI) measured by the Biodex Balance system between the initial assessment and after six weeks of single leg balance training | 6 weeks
  The Overall Stability Index (OASI) is a composite of the Antero-posterior Stability Index (APSI) and the Medio-lateral Stability Index (MLSI)
Assessing change in the time of Single Leg Stance Test between the initial assessment and after six weeks of single leg balance training | 6 weeks
  The time during which the patient is able to stand on one leg measured by seconds

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Ma Elsotohy, Dr, Principal Investigator — Dr
Locations (1):
- Faculty of physical therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anguish B, Sandrey MA. Two 4-Week Balance-Training Programs for Chronic Ankle Instability. J Athl Train. 2018 Jul;53(7):662-671. doi: 10.4085/1062-6050-555-16. PMID 30192681